CLINICAL TRIAL: NCT01089153
Title: Obtaining and Storing Human Blood, Urine, and Fecal Samples for Spirochete-Related Epidemiological Research
Status: Completed | Type: Observational
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Prinicipal Investigator, Southwest Regional Wound Care Center
Other Study IDs: 56-RW-015
Record Dates: First submitted 2010-03-16; First posted 2010-03-18 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: The Samples Will be Studied in Order to Attempt to Better Understand the Occurrence of Blood, Feces and Urine Borne Spirochaetes
Keywords: human blood, urine and fecal samples

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — human blood, urine and fecal samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Current spirochaete infection identification and diagnostic strategies have important limitations. Recent development may allow for an improvement in diagnostic, screening and survey capabilities. The goal of this study is to evaluate blood, urine and fecal samples from a variety of sources and generate information on the occurrence and epidemiology of spirochetes in the general and at risk populations.

DETAILED DESCRIPTION:
The intent of this protocol is to obtain blood, feces and urine samples from subjects with or without a suspected spirochaete infection, so these samples can be used in spirochaete-related scientific studies.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be able to be fully consented to the study.
2. The subject must be 18 years of age or older.
3. The subject must be mentally competent as determined by the Investigator.

Exclusion Criteria:

1. The subject must not be currently incarcerated or pregnant.
2. The subject must not weigh less than 110lbs.
3. If the subject will be contributing more that 60 ml of blood during an 8 (eight) week period, then the subject must not have donated red blood cells within the last 8 (eight) weeks.
4. If the Subject's health would be compromised by contributing up to 30ml of peripheral blood.
5. If in the opinion of the Investigator, the subject has any clinically significant medical diagnosis/conditions which would prevent participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Blood, feces and urine samples may be collected from subjects with known or suspected spirochetal disease or from subjects not suspected to be infected with spirochetes
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Wolcott, MD, Principal Investigator — Southwest Regional Wound Care Center